CLINICAL TRIAL: NCT06025682
Title: Multicenter Retrospective Observational Study Analyzing Infective Complications and the Clinical Outcome of Patients With Acute Lymphoblastic Leukemia Treated With Inotuzumab Ozogamicin (INO-FIRST)
Brief Title: Retrospective Observational Study on Infective Complications and Outcome of Patients With ALL Treated With INO
Acronym: INO-FIRST
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: INF0123
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Acute Lymphoblastic Leukemia; Infections; Bacterial Infections; Viral Infection; Fungal Infection; Acute Lymphoblastic Leukemia, Adult; Acute Lymphoblastic Leukemia, in Relapse
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Infections; Bacterial Infections; Virus Diseases; Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about infectious complications in patients affected by B-cell acute lymphoblastic leukemia treated with inotuzumab-ozogamicin (INO). The main question it aims to answer is:

• incidence of infectious complications (bacterial, fungal, viral) in patients receiving inotuzumab ozogamicin up to 60 days after the end of treatment

DETAILED DESCRIPTION:
The present study is a multicenter, retrospective, observational clinical-epidemiological study on infectious complications (bacterial, fungal, viral) in patients receiving inotuzumab ozogamicin (INO). The study collects data from about 20 Hematologic Centers of the GIMEMA Group treating B-cell acute lymphoblastic leukemia (ALL) patients with inotuzuumab-ozogamicin (INO) over the last 5 years (2018-2023), according to the authorized indications and not included in interventional clinical trials (randomized or not randomized).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Patients with relapsed/refractory CD22 positive B-ALL treated with INO or with relapsed/refractory CD22 positive and Ph-positive B-ALL treated with INO after failing at least one TKI inhibitor
* Signed informed consent if applicable.

Exclusion Criteria:

• Patients treated with INO in interventional clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsed/refractory CD22 positive acute lymphoblastic leukemia treated with INO or with relapsed/refractory CD22 positive and Ph-positive B-ALL treated with INO after failing at least one TKI inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically or microbiologically documented infectious complications in patients receiving inotuzumab ozogamicin (INO) up to 60 days after the end of treatment (last dose administered) | 5 months
  To estimate the rate of clinically or microbiologically documented infectious complications (bacterial, fungal, viral) in acute lymphoblastic leukemia patients receiving inotuzumab ozogamicin (INO) up to 60 days after the end of treatment (last dose administered).

CONTACTS AND LOCATIONS:
Overall Officials: Livio Pagano, Principal Investigator — Policlinico Universitario A. Gemelli, IRCCS-Università Cattolica del Sacro Cuore, Roma
Locations (1):
- UOC Ematologia Fondazione Policlinico Universitario A.Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No